CLINICAL TRIAL: NCT05156424
Title: A Comparison of Aerobic and Resistance Exercise for Counteracting the Adverse Effects of Androgen Deprivation Therapy in Men With Prostate Cancer
Brief Title: A Comparison of Aerobic and Resistance Exercise to Counteract Treatment Side Effects in Men With Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kira Murphy (Other)
Collaborators: Irish Research Council (Other); University of Pittsburgh Medical Center (Other); Waterford Instituate of Technology (Other)
Responsible Party: Sponsor-Investigator, Kira Murphy, Research Coordinator, Waterford Instituate of Technology
Organization: Waterford Instituate of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EBPPG/2020/103
Record Dates: First submitted 2021-10-31; First posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Exercise; Prostate Cancer
Keywords: Prostate Cancer; Physical Fitness; Androgen Deprivation Therapy; Exercise; Cancer
MeSH Terms: conditions — Motor Activity; Prostatic Neoplasms; Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Pilot randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Emphasised Exercise Intervention (Experimental): The intervention will comprise of 24 weeks of twice weekly supervised exercise sessions, emphasising aerobic exercise. To reflect a real-world setting, each group will experience both aerobic and resistance exercise, but there will be a 75%:25% predominant: subsidiary mode emphasis based on exercise duration within each session.
  Interventions: Other: Exercise
- Resistance Emphasised Exercise Intervention (Experimental): The intervention will comprise of 24 weeks of twice weekly supervised exercise sessions, emphasising resistance exercise. To reflect a real-world setting, each group will experience both aerobic and resistance exercise, but there will be a 75%:25% predominant: subsidiary mode emphasis based on exercise duration of exercise within each session.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — An individualised, progressive and autoregulated exercise programme, supervised by a trained professional.

SUMMARY:
Prostate cancer is the second most common cancer in men. Those in the intermediate/high-risk categories typically receive androgen deprivation therapy (ADT) and radiotherapy. ADT greatly reduces androgen production as prostate cancer is dependent on testosterone and dihydrotestosterone for its growth.The side effects of ADT therapy are extensive and include changes in body composition (muscle loss, bone loss and fat gain), strength, mood, physical function, sexual function and increased cardiovascular risk and fatigue. Many of these side effects can be influenced by exercise training, both resistance training and aerobic training. However, the most appropriate exercise regime for men undergoing ADT has received little research attention.

DETAILED DESCRIPTION:
Although many interventions for prostate survivors emphasise resistance exercise to maintain muscle mass and strength. Arguments could equally be made for programmes emphasising aerobic exercise for fatigue, anxiety, cardiovascular risk reduction and indeed overall survival.

Comparisons of programmes that emphasise each exercise mode are clearly required.

Therefore the overall purpose of this feasibility and pilot randomised control trial is to determine the feasibility and preliminary effectiveness of an aerobic emphasised exercise program (AE) verses a resistance emphasise exercise program (RE) in a rehabilitation setting, over 6 months, for prostate cancer men undergoing Androgen Deprivation Therapy (ADT).

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age with a histologically diagnosed prostate cancer
* Prescribed ADT (Androgen deprivation Therapy)
* Self-reported not to be partaking in regular exercise (structured aerobic or resistance training ≥ 2 sessions/week) in the past 3 months.
* Medically cleared to exercise by their oncologist

Exclusion Criteria:

* Prior exposure to ADT >12 months
* Prior hypogonadism
* Established metastatic bone disease
* Established Osteoporosis
* Musculoskeletal/Cardiovascular and/or Neurological disease that could put them at risk from exercise as judged by the attending physician.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men diagnosed with prostate cancer will be recruited.
Enrollment: 24 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility- recruitment rate (%) | At study conclusion
  The recruitment rate will be established by comparing the number of potential participants approached and how many agreed to participate in the trial. This will be reported in percentage format.
Feasibility- retention rate (%) | Intervention conclusion 24 weeks
  Percentage of participants that completed the 24 week intervention compared to the number of participants randomised. This will be reported in percentage format.
Feasibility- exercise program adherence through attendance %. | Throughout 24 week intervention
  The research team will report adherence to the exercise program through attendance of supervised classes. Attendance will be reported as a percentage.
Feasibility- exercise prescription adherence (% of modified sessions compared to attended exercise sessions) | Throughout 24 week intervention
  The research team will report adherence to the exercise prescription by reporting the number of modified sessions compared to attended exercise sessions. This will be reported as a percentage.
Feasibility- Adverse Event using CTCAE v4.0 grading system. | At study conclusion
  The research team will report any adverse events in general or in relation to the exercise program using CTCAE v4.0 grading system.
Feasibility- Patient satisfaction/acceptability through qualitative evaluation. | Following intervention conclusion at 24 weeks
  Determined by qualitative evaluation, using semi structured interviews and exit surveys to evaluate the acceptability, experiences and feasibility of the intervention.

SECONDARY OUTCOMES:
General quality of life by questionnaire | At baseline, 8 weeks and 24 weeks (end of intervention)
  The RAND 36-Item Health Survey comprises of 36 questions and assesses eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scores range from 0-100. A higher score indicates a high quality of life and a favourable health status.
Cancer Specific quality of life by questionnaire | At baseline, 8 weeks and 24 weeks (end of intervention)
  The European Organisation for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) comprises of 30 questions, categorised into five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item (dyspnoea, appetite loss, sleep disturbance, constipation, diarrhoea and the financial impact) scales assess symptoms.
  Scores range from 0-100. A higher score for the functional scales and global health status indicates better functioning and quality of life. A higher score on the symptom and single-item scales denotes a high level of symptoms (i.e. a poor quality of life).
Prostate cancer specific quality of life by questionnaire | At baseline, 8 weeks and 24 weeks (end of intervention)
  The European Organisation for the Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-PR25) is a prostate cancer supplementary questionnaire module to be employed in conjunction with EORTC QLQ-C30. It comprises of five multi-item scales to assess sexual activity, sexual functioning, urinary symptoms, bowel symptoms and hormonal treatment-related symptoms and one single item assessing incontinence. Scores range from 0-100. A high score for the sexual activity and sexual functioning scales represents a high level of functioning. A high score for urinary, bowel and hormonal treatment related symptoms scales and incontinence aid item represents a high level of symptomatology.
Fatigue by questionnaire | At baseline, 8 weeks and 24 weeks (end of intervention)
  The Functional Assessment of Cancer Therapy - Fatigue (FACIT-Fatigue) questionnaire will be used to measure fatigue. Patients will score 13 fatigue items over the past 7 days on a scale (0 = not at all; 4 = very much), generating a total (0 - 52). A higher score indicates lower levels of fatigue.
Physical Activity (subjective) by questionnaire | At baseline, 8 weeks and 24 weeks (end of intervention)
  The Godin Leisure Time Exercise questionnaire will be used to calculate the average amount of strenuous, moderate and light exercise a participant performs in a typical 7 day period. A score of 24 units or more indicates the participant is active, 14-23 units indicates moderately active and less than 14 units suggests the participant is insufficiently active/sedentary.
Anthropometric assessment. | At baseline and 24 weeks (end of intervention)
  Height will be measured in cm and body weight in kg, which will be combined to report BMI in kg/m(squared).
Waist and Hip circumference analysis (cms) | At baseline and 24 weeks (end of intervention)
  Waist circumference and hip circumference will be measured in centimetres. These two measurements will be used to calculate the participants waist: hip ratio. All measurements will be taken in duplication and averaged before data entry. If there is a substantial difference between the two measures, a third measurement will be taken.
Body composition (fat mass) analysis using Dual Energy X Ray Absorptiometry (Dexa) | At baseline and 24 weeks (end of intervention)
  Fat mass (grams and percentage) will be assessed using DEXA (Horizon W, Hologic, 304492M). Participants will be scanned after an overnight fast and will be instructed to regulate their water/fluid intake in the days leading up to the scan, so they are adequately hydrated. All scans will be completed at the same time as much as possible to account for physiological changes in body composition throughout the day.
Body composition (fat and lean mass) analysis using Dual Energy X Ray Absorptiometry (Dexa) | At baseline and 24 weeks (end of intervention)
  Lean mass (grams and percentage) will be assessed using DEXA (Horizon W, Hologic, 304492M). Participants will be scanned after an overnight fast and will be instructed to regulate their water/fluid intake in the days leading up to the scan, so they are adequately hydrated. All scans will be completed at the same time as much as possible to account for physiological changes in body composition throughout the day.
Bone density (BMD) measurement | At baseline and 24 weeks (end of intervention)
  Whole body bone Density will be measured using DEXA (Horizon W, Hologic, 304492M). BMD will be measured in g/cm(squared) and used to calculate a T-score (SD). A T-score shows how much a participant's BMD is higher or lower than the BMD of a healthy 30 year old adult and is the score most commonly used to diagnose low BMD.
Visceral fat area (VAT Area) in cm(squared) | At baseline and 24 weeks (end of intervention)
  Visceral fat area will be assessed using DEXA (Horizon W, Hologic, 304492M). It will be measured in cm(squared). Participants will be scanned after an overnight fast and will be instructed to regulate their water/fluid intake in the days leading up to the scan, so they are adequately hydrated. All scans will be completed at the same time as much as possible to account for physiological changes in body composition throughout the day
Atrial stiffness measured by a Pulse Wave Velocity Assessment (m/s) | At baseline and 24 weeks (end of intervention)
  A carotid-femoral pulse wave velocity test will be performed to assess arterial stiffness. It will be measured in meters per seconds (m/s). This will be performed as per manufactural instructions using a Complior, Alam medical device. Measurements will be taken in duplicate and the mean recorded, with a third measurement taken if difference between the two measurements is more than 0.5 m/s and median recorded.
Blood pressure (mmHg) | At baseline and 24 weeks (end of intervention)
  Blood pressure (diastolic and systolic) measured at rest. Blood pressure will be taken according to the American Heart Association's (AHA) guidelines. At least two readings and the average recorded. Additional readings will be taken if the difference between the two reading exceeds 5mm Hg.
Cardiovascular Fitness | 0(baseline), 8 weeks and 6 months (end of intervention)
  Cardiovascular fitness will be determined by a submaximal incremental treadmill test using a modified Bruce protocol. The test will be scored by the time (minutes and seconds) taken to test completion. A longer time to completion means superior cardiovascular fitness.
Peak torque/power for knee extension and flexion | At baseline and 24 weeks (end of intervention)
  An isokinetic dynamometry for knee extension and flexion will also be performed on a Biodex (Advantage BX™ Software Update v5.3.00) to measure peak torque (n.M) and power, using a similar protocol as previously used in cancer patients.
Lower limb strength [Leg Press] | At baseline and 24 weeks (end of intervention)
  Leg press 1 repetition maximum will be measured in kilograms (kg). A 1 repetition maximum is defined as the highest load that can be lifted through full range of movement for one time.
Upper limb strength [Chest Press] | At baseline and 24 weeks (end of intervention)
  Chest press 1 repetition maximum will be measured in kilograms (kg). A 1 repetition maximum is defined as the highest load that can be lifted through full range of movement for one time.
Functional Ability Assessment (Timed up and go) | At baseline, 8 weeks and 24 weeks (end of intervention)
  The timed up and go assess the time (in seconds) it takes for a person to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees. It assesses mobility, balance, walking ability and falls risk in older adults. A lower score indicates better physical function.
Functional Ability Assessment (Sit to stand) | At baseline, 8 weeks and 24 weeks (end of intervention)
  Sit to stand assesses the maximal repetitions a participant can stand up from a chair in 30 seconds. A higher score indicates better physical function.
Functional Ability Assessment (Grip test) | At baseline, 8 weeks and 24 weeks (end of intervention)
  A hand-held dynamometry will be used to measure grip strength for each arm. this is a measure of upper body strength and a higher score suggests better upper body strength
Functional Ability Assessment (Bess Balance test) | At baseline, 8 weeks and 24 weeks (end of intervention)
  The Balance Error Scoring System is an objective measure of assessing static postural stability. A lower score= better balance and reduced falls risk.
Functional Ability Assessment (6 minute walk test) | At baseline, 8 weeks and 24 weeks (end of intervention)
  A 6-min walk test measured the maximal meters walked in six minutes. A higher score indicated superior aerobic endurance and capacity.
Functional Ability Assessment (Sit and reach) | At baseline, 8 weeks and 24 weeks (end of intervention)
  The sit and reach test measures linear flexibility. The score is the most distant point (cm) reached with the fingertips. A higher score indicates better flexibility
Biomarker Analysis: Blood lipids (mmol/L) | At baseline and 24 weeks (end of intervention)
  Blood lipids (total cholesterol, triglycerides, LDH and HDL) will be analysed Fasting blood will be taken from all participants using a standard venipuncture technique. All bloods will be analyzed in a certified clinical lab.
Biomarker Analysis: Glucose (mmol/L) | At baseline and 24 weeks (end of intervention)
  Fasted blood will be used to measure blood glucose (mmol/L),
Biomarker Analysis: Insulin (mIU/L) | At baseline and 24 weeks (end of intervention)
  Fasted blood will be used to measure blood insulin (mIU/L)
Biomarker Analysis: C-Reactive Protein (CRP) | At baseline and 24 weeks (end of intervention)
  Fasted blood will be used to measure C-reactive protein (mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dr Harrison, PhD, Principal Investigator — Waterford Institute of Technology
Locations (1):
- WIT Sports Arena, Waterford, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cancer statistics. Viewed 21st February 2020. https://www.cancer.ie/cancer-information-and-support/cancer-information/about-cancer/cancer-statistics
- [Background] Hormone Therapy for Prostate Cancer. Viewed on the 20th January 2020 https://www.cancer.org/cancer/prostate-cancer/treating/hormone-therapy.html
- [Background] Bylow K, Mohile SG, Stadler WM, Dale W. Does androgen-deprivation therapy accelerate the development of frailty in older men with prostate cancer?: a conceptual review. Cancer. 2007 Dec 15;110(12):2604-13. doi: 10.1002/cncr.23084. PMID 17960609
- [Background] Norris MK, Bell GJ, North S, Courneya KS. Effects of resistance training frequency on physical functioning and quality of life in prostate cancer survivors: a pilot randomized controlled trial. Prostate Cancer Prostatic Dis. 2015 Sep;18(3):281-7. doi: 10.1038/pcan.2015.28. Epub 2015 Jun 16. PMID 26078203
- [Background] Fairman CM, Kendall KL, Hart NH, Taaffe DR, Galvao DA, Newton RU. The potential therapeutic effects of creatine supplementation on body composition and muscle function in cancer. Crit Rev Oncol Hematol. 2019 Jan;133:46-57. doi: 10.1016/j.critrevonc.2018.11.003. Epub 2018 Nov 12. PMID 30661658
- [Background] Winters-Stone KM, Lyons KS, Dobek J, Dieckmann NF, Bennett JA, Nail L, Beer TM. Benefits of partnered strength training for prostate cancer survivors and spouses: results from a randomized controlled trial of the Exercising Together project. J Cancer Surviv. 2016 Aug;10(4):633-44. doi: 10.1007/s11764-015-0509-0. Epub 2015 Dec 29. PMID 26715587
- [Background] Nilsen TS, Raastad T, Skovlund E, Courneya KS, Langberg CW, Lilleby W, Fossa SD, Thorsen L. Effects of strength training on body composition, physical functioning, and quality of life in prostate cancer patients during androgen deprivation therapy. Acta Oncol. 2015 Nov;54(10):1805-13. doi: 10.3109/0284186X.2015.1037008. Epub 2015 Apr 30. PMID 25927504
- [Background] Newton RU, Kenfield SA, Hart NH, Chan JM, Courneya KS, Catto J, Finn SP, Greenwood R, Hughes DC, Mucci L, Plymate SR, Praet SFE, Guinan EM, Van Blarigan EL, Casey O, Buzza M, Gledhill S, Zhang L, Galvao DA, Ryan CJ, Saad F. Intense Exercise for Survival among Men with Metastatic Castrate-Resistant Prostate Cancer (INTERVAL-GAP4): a multicentre, randomised, controlled phase III study protocol. BMJ Open. 2018 May 14;8(5):e022899. doi: 10.1136/bmjopen-2018-022899. PMID 29764892
- [Background] Kilgour RD, Vigano A, Trutschnigg B, Hornby L, Lucar E, Bacon SL, Morais JA. Cancer-related fatigue: the impact of skeletal muscle mass and strength in patients with advanced cancer. J Cachexia Sarcopenia Muscle. 2010 Dec;1(2):177-185. doi: 10.1007/s13539-010-0016-0. Epub 2010 Dec 17. PMID 21475694
- [Background] Van Bortel LM, Laurent S, Boutouyrie P, Chowienczyk P, Cruickshank JK, De Backer T, Filipovsky J, Huybrechts S, Mattace-Raso FU, Protogerou AD, Schillaci G, Segers P, Vermeersch S, Weber T; Artery Society; European Society of Hypertension Working Group on Vascular Structure and Function; European Network for Noninvasive Investigation of Large Arteries. Expert consensus document on the measurement of aortic stiffness in daily practice using carotid-femoral pulse wave velocity. J Hypertens. 2012 Mar;30(3):445-8. doi: 10.1097/HJH.0b013e32834fa8b0. PMID 22278144
- [Background] Flack JM, Adekola B. Blood pressure and the new ACC/AHA hypertension guidelines. Trends Cardiovasc Med. 2020 Apr;30(3):160-164. doi: 10.1016/j.tcm.2019.05.003. Epub 2019 May 15. PMID 31521481
- [Derived] Murphy K, Kehoe B, Denieffe S, Hacking D, Fairman CM, Harrison M. Comparing aerobic and resistance exercise emphasis during androgen deprivation and radiation therapy for prostate cancer: A randomised feasibility trial. Support Care Cancer. 2025 Jun 20;33(7):601. doi: 10.1007/s00520-025-09650-z. PMID 40540036
- [Derived] Murphy K, Kehoe B, Denieffe S, McGrath A, Hacking D, Fairman CM, Harrison M. 'Just because I have prostate cancer doesn't mean that I can't do things' - men's experiences of the acceptability of an exercise intervention for prostate cancer during treatment. BMC Cancer. 2024 Aug 2;24(1):949. doi: 10.1186/s12885-024-12687-8. PMID 39095735